CLINICAL TRIAL: NCT01071681
Title: Observational Survey Assessing the Factors of Treatment Intensification in Uncontrolled Hypertensive Patients Under a Combination Therapy, Either Fixed or Not, of a Renin-Angiotensin System Blocker (RASB) and Hydrochlorothiazide (HCTZ), According to Their Level of Cardiovascular Risk.
Brief Title: Survey to Assess Why People Are Not Responding to Treatment in Hypertension
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: International Clinical Trials Association (Other)
Responsible Party: Medical Director, Bayer Schering Pharma AG
Other Study IDs: 14675; KL0911FR (Other: Company Internal); BI INTENS (Other: Company Internal)
Record Dates: First submitted 2009-10-01; First posted 2010-02-19 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Arterial Hypertension
Keywords: Arterial hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Telmisartan (Kinzal/Pritor, BAY68-9291)

INTERVENTIONS:
Drug: Telmisartan (Kinzal/Pritor, BAY68-9291) — Patients under daily life treatment receiving Pritor according to local drug information.

SUMMARY:
This study will describe the factors influencing the physician in face of elevated blood pressure in already treated patients

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18
* Hypertensive patients
* Uncontrolled hypertension (blood pressure >/=140/90 mmHg on the day of consultation or >/=130/80 mmHg in diabetic patients or in patients suffering from kidney failure, or in elderly patients with a systolic blood pressure >/=150 mmHg (in the absence of orthostatic hypotension)
* Patients treated with a combination, fixed or not, of Renin-Angiotensin System Blocker (RASB) + Hydrochlorothiazide (HCTZ)
* Patients examined in common medical care practice, whatever the reason for consultation
* Patients informed of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Uncontrolled hypertensive patients under a combination therapy, either fixed or not, of a renin-angiotensin system blocker and hydrochlorothiazide
Sampling Method: Non-Probability Sample
Enrollment: 1589 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients, according to the level of cardiovascular risk, who, at the end of the visit:- do not present any modification of hypertension treatment (therapeutic inertia) - present a change in the hypertension therapeutic | on day 1

SECONDARY OUTCOMES:
Analyses of the factors that had an impact on the therapeutic decision | on day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, France